CLINICAL TRIAL: NCT01494974
Title: Comparison of the Ahmed Glaucoma Valve FP7 and FP8 in Pediatric Glaucoma: a Randomized Clinical Trial.
Brief Title: Comparison of the Ahmed Glaucoma Valve FP7 and FP8 in Pediatric Glaucoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Camila Fonseca Netto, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 0236/11
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Pediatric Glaucoma
Keywords: Glaucoma; Pediatric; Ahmed; Congenital; FP7; FP8
MeSH Terms: conditions — Hydrophthalmos; Glaucoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FP7 implant (Active Comparator)
  Interventions: Device: FP7 Ahmed Glaucoma Drainage Implant
- FP8 implant (Active Comparator)
  Interventions: Device: FP8 Glaucoma Drainage Implant

INTERVENTIONS:
Device: FP7 Ahmed Glaucoma Drainage Implant — Ahmed Glaucoma Valve model FP7
  Arms: FP7 implant
Device: FP8 Glaucoma Drainage Implant — Ahmed Glaucoma Valve model FP8
  Arms: FP8 implant

SUMMARY:
The purpose of this study is to compare the success rates and complications of two models of Ahmed glaucoma implants (FP7 and FP8) in patients with pediatric glaucoma.

DETAILED DESCRIPTION:
INTRODUCTION

The drainage implants have become an important alternative in the treatment of pediatric glaucoma refractory to angular and filtration surgery or medical therapy (1). Such implants drain the aqueous humor from the anterior chamber of the eye to a plate positioned above the sclera, between the rectus muscles. The aqueous humor goes through the pseudocyst that forms around the plate by passive diffusion and is drained by the venous capillaries and lymphatic system.

The Ahmed drainage implant (New World Medical, Inc., Rancho Cucamonga, CA, USA) is a device with flow restrictors, which decreases the incidence of postoperative complications such as hypotony (2-3). It is made of silicone and comes in two sizes. The FP7 model has a surface of 184 mm2, 13mm wide and 16mm long. The FP8 model presents 96mm2 surface, 9.6 mm wide and 10mm long.

Studies in animals and adult humans suggest that the surface area of the implant plate is directly related to the amount of aqueous fluid drained through the same (4-7). In contrast, a very large implant can result in the extrusion of the same, uncontrolled intraocular pressure, corneal injury by endothelial touch, patient discomfort and ocular motility problems. The use of pediatric size implants in small eyes can avoid such complications. A high rate (34.8%) of anterior plate of the tubes in children under 2 years of age has been reported (8-9). On the other hand, the use of pediatric implante may affect the control of intraocular pressure (IOP) due to reduced drainage area (10), especially in eyes with increasing axial diameter, a result of increased eye pressure that happens in children with glaucoma. However, there is no study in the literature comparing different sizes of drainage implants in pediatric patients.

A study to compare the success rates and complications between FP7 and FP8 models is essential in order to standardize a conduct in choosing the type of implant. Currently, the choice of the drainage implant model to be used in every child lies on the free choice and personal preference of the surgeon. There is no standard procedure, based on scientific evidence for this choice.

OBJECTIVES

Compare the success rates and complications of two models of Ahmed drainage implant (FP7 and FP8) in patients with pediatric glaucoma.

MATERIALS AND METHODS

This clinical trial is a prospective, randomized, masked to the evaluator to be held at the Department of Ophthalmology, Federal University of Sao Paulo.

Will be included children between 0 and 10 years of age with glaucoma and surgical indication for glaucoma drainage implant. Surgical indication for implantation of Ahmed drainage occurs in some situations: 1) children with primary congenital glaucoma that undergone angular surgery (goniotomy and / or trabeculotomy) who did not respond satisfactorily to surgery, 2) children with glaucoma secondary to aphakia who have the primary indication for implantation of Ahmed drainage, 3) children with glaucoma secondary to other eye disorders where medical treatment is not satisfactory.

A term of consent will be obtained from parents or legal guardians of the child, in which all the risks inherent to the surgical procedure will be clarified. Such risks are proper to antiglaucomatous surgery are:

1. Early: hypotony, hyphema, tube endothelial touch, choroidal detachment, leakage of aqueous, vitreous hemorrhage, retinal detachment, loss of light perception
2. late: uncontrolled intraocular pressure, persistent hypotony, scleral patch resorption, extrusion of the tube, retinal detachment, loss of light perception (11-18).

Considering that the selected patient has already the surgical indication for Ahmed drainage implant, the inclusion of this child in the study does not bring additional risks or discomforts to the same.

The model of the drainage implant will be chosen through allocation from a computer-generated random table.

Children enrolled in the study will be divided into two groups (one group will receive the model FP7 and another group will receive the model FP8) with the number of 20 participants in each group, totaling 40 children.

The surgeries will be performed by experienced surgeons from Glaucoma Sector from Department of Ophthalmology, Federal University of Sao Paulo.

The plate of the Ahmed drainage implant will be placed in one of the quadrants selected from the extraocular muscles between 8 and 10 mm away from the corneal limbus. The tube will have its distal portion inserted 2-3mm into the anterior chamber of the eye in the iris plane. The exposed portion of the tube is covered with donor sclera.

The children included in the study will be examined before surgery, which will be measured your visual acuity, biomicroscopy, IOP, Retinography and axial length of the eye. Immediately after surgery, with a compass we will measure the distance between the plate of drainage implant and corneal limbus.

Children will be examined again after 6 months and 1 year of surgery. We will perform the measurement of visual acuity, biomicroscopy, IOP, Retinography, axial length and measurement of the distance from the plate of the implant and corneal limbus. Post-operative examinations will be performed under narcosis, in hospitals (when it is impossible to take measures in an outpatient setting due to lack of cooperation of the child), by a doctor from congenital glaucoma sector who were not involved in the surgical procedure. The examination under narcosis involves risk to the child, which include cough, nausea, vomiting, laryngospasm, bronchospasm, apnea, bradycardia, tachycardia, hypertension, anxiety (19-21).

Two types of outcome will be considered in this study. The primary endpoint is to evaluate the position of the drainage implant plate and if the plate is positioned at a distance ≥ 8 mm from the corneal limbus after 1 year of surgery, considered successful. If the dish drain implant is positioned at a distance <8 mm from the corneal limbus, we have a failure.

As a secondary outcome, we evaluate the variation in IOP preoperative and postoperative. We will use as a criterion of success an IOP ≤ 21 mm Hg and> 5 mmHg and a 30% reduction of preoperative IOP. If the patient meets these criteria, without the use of eyedrop, classified as complete success. If the use of eyedrop is necessary to meet the criteria, a qualified success will be defined.

For failure criterion is assumed: IOP ≤ 5 mmHg or > 21 mm Hg, even with the use of eye drops, need for further surgery, and / or loss of light perception.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Pediatric Glaucoma with indication of Ahmed Glaucoma Valve implantation
* Age from 0 to 10 years old

Exclusion Criteria:

* Children older then 10 years old

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Position of the drainage implant plate | After 1 year of surgery
  The primary endpoint is to evaluate the position of the drainage implant plate and if the plate is positioned at a distance ≥ 8 mm from the corneal limbus after 1 year of surgery, considered successful. If the plate is positioned at a distance <8 mm from the corneal limbus, we have a failure.

SECONDARY OUTCOMES:
As a secondary outcome, we evaluate the variation in IOP preoperative and postoperative. | After 1 year of surgery
  We will use as a criterion of success an IOP ≤ 21 mm Hg and> 5 mmHg and a 30% reduction of preoperative IOP. If the patient meets these criteria, without the use of eyedrop, classified as complete success. If the use of eyedrop is necessary to meet the criteria, a qualified success will be defined.
  For failure criterion is assumed: IOP ≤ 5 mmHg or > 21 mm Hg, even with the use of eye drops, need for further surgery, and / or loss of light perception.

CONTACTS AND LOCATIONS:
Overall Officials: Camila F Netto, MD, Principal Investigator — Assistant Doctor at Ophthalmology Department
Locations (1):
- Federal University of São Paulo - Ophthalmology Department, São Paulo, São Paulo, Brazil